CLINICAL TRIAL: NCT04098497
Title: Modeling Mood Course to Detect Markers for Effective Adaptive Interventions- Aim 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1322 Aim-3; Biostat & Med (Other: UW, Madison); 7K01MH112876-02 (NIH); A538500 (Other: UW Madison); SMPH/POP HEALTH SCI/POP HEALTH (Other: UW Madison)
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Bipolar Disorder; Psychosocial Intervention
Keywords: mood; stress; sleep; circadian rhythm; medical adherence; acceptance and commitment therapy; microintervention
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This study uses a design known as a microrandomized trial. Whereas a multi-arm trial randomizes a subject to an intervention group only once at the start of the study, a microrandomized trial repeatedly randomizes a subject to an intervention group throughout the study. In addition to an overall effect of an intervention on proximal outcomes, a microrandomized trial allows one to determine if the effect is modified by momentary factors (e.g., current mood, day of the week, day in the study).
  For the present study, every subject has a equal chance of being assigned to one of two intervention groups at each of 84 time points (2 daily x 42 days). At each time point, the two intervention groups are to either receive a prompt based on Acceptance and Commitment Therapy (ACT) or not receive such a prompt. Regardless of the assigned group, subjects are asked to assess their mood, stress, and activity at every time point prior to assignment to intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-based microintervention delivered by mobile app (Experimental): At every time-point of the study, participants will complete self-reports of mania (as measured by the shortened YMRS), depression (as measured by the shortened SIGH-D ), medication adherence, and activity through the mobile app Lorevimo. After completing these assessments, participants will be randomly assigned to either receive one additional ACT-based microintervention question or receive no additional question.
  The microintervention will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT (contacting the present moment, defusion, acceptance, self-as-context, values, and committed action).
  The ACT-based questions were developed by the research team as a unique intervention for the current study. They are based upon core themes of acceptance and commitment therapy: engagement, awareness, and openness.
  Interventions: Behavioral: Mobile intervention

INTERVENTIONS:
Behavioral: Mobile intervention — The mobile intervention in this study consists of two components: 1) self-monitoring and 2) an ACT-based microintervention.
  Self-monitoring: twice daily, participants will complete self-reports of mania, depression, medication adherence, and activity through the mobile app Lorevimo.
  Microintervention: The microintervention will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT (contacting the present moment, defusion, acceptance, self-as-context, values, and committed action). At each time-point, participants have a 50% chance of receiving a microintervention question along with the daily self-monitoring assessments.

SUMMARY:
This study is a 6-week micro-randomized trial investigating the feasibility of a mobile health platform. Its long-term objective is to develop a mobile health platform for the translation of a psychosocial intervention for bipolar disorder (BP) into an effective and evidence-based adaptive intervention. In this aim of the study, investigators will evaluate how individuals with BP respond to a microintervention based in acceptance and commitment therapy (ACT) that is delivered with a mobile app.

DETAILED DESCRIPTION:
Bipolar (BP) disorder is a chronic illness of profound shifts in mood ranging from mania to depression. BP is successfully treated by combining medication with psychosocial therapy, but care can prove inadequate in practice. With gaps in coverage and medication, along with imprecise guidelines on when, where, and how to intervene, promising psychosocial therapies require adaptive strategies to better address the specific needs of individuals in a timely manner. However, To accomplish this, evidence based practices are needed. This project aims to address this knowledge gap by establishing a mobile health platform for translating a psychosocial therapy in BP into an effective adaptive intervention.

The research to be conducted under this protocol falls under the general heading of a micro-randomized trial. It investigates feasibility of a study on how to tailor an intervention based on acceptance and commitment therapy (ACT) when delivered via a smartphone app. Long-term objective of this study is to develop a mobile health platform for the translation of a psychosocial intervention for bipolar disorder (BP) into an effective adaptive intervention. In this particular part of the study, the investigator will assess the feasibility of a mobile health and wearable device platform for the translation of a BP psychosocial therapy into an evidenced-based adaptive intervention. To answer this question, investigator will study how individuals with BP respond to a microintervention delivered via a mobile app. Primary outcome of this study is to evaluate the feasibility of a micro-randomized trial in ACT in terms of completion of assessments (interview and self-report), wearing of Fitbit, and completion of microintervention questions. Secondary outcome of the study is to detect a linear effect in time of the microintervention on symptom levels of mania and depression in individuals with bipolar disorder. The estimated linear effect would be used to power a larger study.Enrollment is by invitation only; participants in the study will be recruited from the Prechter Longitudinal Study of Bipolar Disorder (HUM606).

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Bipolar Disorder
* have agreed to be contacted for future research
* have a smart-phone
* have a diagnosis of bipolar disorder.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melvis Mclnnis, MD, Principal Investigator — University of Michigan, Ann Arbor, MI
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cochran A, Maronge JM, Victory A, Hoel S, McInnis MG, Thomas EB. Mobile Acceptance and Commitment Therapy in Bipolar Disorder: Microrandomized Trial. JMIR Ment Health. 2023 Apr 20;10:e43164. doi: 10.2196/43164. PMID 37079363
- [Derived] Kroska EB, Hoel S, Victory A, Murphy SA, McInnis MG, Stowe ZN, Cochran A. Optimizing an Acceptance and Commitment Therapy Microintervention Via a Mobile App With Two Cohorts: Protocol for Micro-Randomized Trials. JMIR Res Protoc. 2020 Sep 23;9(9):e17086. doi: 10.2196/17086. PMID 32965227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Milestones are not mutually exclusive; e.g., one participant could complete the exit interview, but never set up the Fitbit. All participants were included in at least one component of the analysis. The one participant who did not complete the final interview was not included in the analysis of safety outcomes. The four participants who were never randomized were not included in the analysis of effectiveness outcomes. All participants were included in the analysis of feasibility outcomes.
Pre-assignment Details: Participants were recruited from a longitudinal cohort of bipolar disorder, so initial screening was not needed
Groups:
- ACT-based Microintervention Delivered by Mobile App: The ACT-based questions were developed by the research team as a unique intervention for the current study. They are based upon core themes of acceptance and commitment therapy: engagement, awareness, and openness.
  Mobile intervention: The mobile intervention in this study consists of two components: 1) self-monitoring and 2) an ACT-based microintervention.
  Self-monitoring: twice daily, participants will complete self-reports of mania, depression, medication adherence, and activity through the mobile app Lorevimo.
  Microintervention: The microintervention will consist of one of 84 prompts that aim to target one of 6 processes targeted in ACT (contacting the present moment, defusion, acceptance, self-as-context, values, and committed action). At each time-point, participants have a 50% chance of receiving a microintervention question along with the daily self-monitoring assessments.
Period: Overall Study
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Started | 30
Initial Interview | 30
Set Up Study App | 29
Logged Symptoms Into Study App at Least Once (Participants who did not log symptoms into the app were never randomized to receive or not receive an intervention) | 26
Linked Fitbit to Study Database | 27
Used Fitbit | 24
Exit Interview (Participant who did not do the exit interview was not included in analysis of safety outcomes.) | 29
Completed (All participants were included in the analysis of feasibility outcomes) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.70 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 25
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Diagnosis [Count of Participants; unit: Participants] — Bipolar I = history of mania Bipolar II = history of depression and hypomania Bipolar NOS = Not Otherwise Specified, suggestive of Bipolar disorder, but not indicative
  Participants
    Bipolar I | 24
    Bipolar II | 6
    Bipolar NOS | 0
Baseline HRSD Score [Mean (Standard Deviation); unit: score on a scale] — Hamilton Depression Rating Scale (HDRS), scores range from 0-54 with higher scores indicating increased depression.
  score on a scale | 6.20 (5.78)
Baseline YMRS Score [Mean (Standard Deviation); unit: score on a scale] — Young Mania Rating Scale (YMRS) Scores range from 0-60 with higher scores indicative of increased mania
  score on a scale | 1.83 (3.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Shortened YMRS Surveys Completed
Description: Feasibility of the microintervention will be evaluated by measuring the average completion of the shortened Young Mania Rating Scale (YMRS) that will be delivered to participants through the mobile app. Number of completed surveys is reported.
  The Young Mania Rating Scale (YMRS) is a 11-item interview-based measure of manic symptoms. Scores on 3 items range from 0 to 8, whereas scores on the remaining 8 items range from 0 to 4. The total score of the YMRS can range from 0 to 60, with higher scores indicating more severe manic symptoms.
  The shortened scale used for the app includes three items (tracking the symptoms increased energy, rapid speech, and irritability) from the YMRS. The symptoms are scored on the following 0-3 scale:
  0 = absent/normal
  1. = mild
  2. = moderate
  3. = severe
Time Frame: Days 1-43
Population: All participants were included in the analysis of feasibility outcomes. 30 participants were planned to receive 84 decision points for a total possible number of 2520 surveys delivered.
Measure: Number; unit: completed surveys
Units Other Than Participants: surveys delivered
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 30
Number analyzed (surveys delivered) | 2520
completed surveys | 1651

2. Primary Outcome: Number of Shortened SIGHD Surveys Completed
Description: Feasibility of the microintervention will be evaluated using the average completion of the shortened Structured Interview Guide for the Hamilton Depression Rating Scale (SIGH-D) that will be delivered to participants through the mobile app. Number of completed surveys is reported.
  The SIGH-D is a 17-item clinician-rated scale that assesses the severity of depressive symptoms. The total score is obtained by summing the score of each item, 0-4 (symptom is absent, mild, moderate, or severe) or 0-2 (absent, slight or trivial, clearly present). Scores can range from 0 to 54, with higher scores indicating more severe depression.
  The shortened SIGH-D assessment contains three items that track symptoms of depressed mood, fidgeting, and fatigue. The symptoms are scored on the following 0-3 scale:
  0 = absent/normal
  1. = mild
  2. = moderate
  3. = severe
Time Frame: Days 1-43
Population: as for outcome 1
Measure: Number; unit: completed surveys
Units Other Than Participants: surveys delivered
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 30
Number analyzed (surveys delivered) | 2520
completed surveys | 1651

3. Primary Outcome: Change in YMRS Score
Description: The safety of the microintervention will be assessed by examining the change in YMRS scores from the beginning of the study (YMRS administered in entrance interview) to the end (YMRS administered again in exit interview).
  The Young Mania Rating Scale (YMRS) is a 11-item interview-based measure of manic symptoms. Scores on 3 items range from 0 to 8, whereas scores on the remaining 8 items range from 0 to 4. The total score of the YMRS can range from 0 to 56, with higher scores indicating more severe manic symptoms.
Time Frame: Day 0, Day 42
Population: One participant did not complete the Exit Interview and therefore safety data is not available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 29
score on a scale | -1.2 (3.75)
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; baseline to day 42 comparison; Test type: Other; p = 0.09, t-test, 2 sided; t = 1.74, df = 28

4. Primary Outcome: Change in SIGH-D Score
Description: The safety of the microintervention will be assessed by examining the change in SIGH-D scores from the beginning of the study (SIGH-D administered in entrance interview) to the end (SIGH-D administered again in exit interview).
  The SIGH-D is a 17-item clinician-rated scale that assesses the severity of depressive symptoms. The total score is obtained by summing the score of each item, 0-4 (symptom is absent, mild, moderate, or severe) or 0-2 (absent, slight or trivial, clearly present). Scores can range from 0 to 54, with higher scores indicating more severe depression.
Time Frame: Day 0, Day 42
Population: One participant did not complete the Exit Interview and therefore safety data is not available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 29
score on a scale | 2.1 (6.59)
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; baseline to day 42; Test type: Other; p = 0.09, t-test, 2 sided; t = 1.75, df = 28

5. Secondary Outcome: Average Change in m Score on digiBP From One Decision Time Point to the Next Decision Time Point as a Result of the Intervention
Description: Mood was self-reported using the 6-item digital survey for mood in bipolar disorder (digiPB). This survey is comprised of 3 items (depressed mood, fatigue, fidgeting) measuring common depressive symptoms, two items (increased energy, rapid speech) measuring common manic symptoms, and one item (irritability) measuring a common symptom of both mania and depression. Each item is rated on ordinal scale: 0=absent/normal, 1=mild, 2=moderate, 3=severe. Two scores, d and m, are computed to measure severity of depressive and manic symptoms, respectively. The m score ranges from 0 to 18 with higher scores being most severe symptoms of mania. Self-reported mood was collected twice-daily over 42 days, once in the morning and once in the evening. This leads to a total of 84 decision time points. This outcome looks at the average change in the m score from one decision time point to the next (e.g., from morning to evening or from evening to the next morning) that is attributed to the intervention.
Time Frame: data collected twice daily over 42 days (Days 1-43)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 26
score on a scale | 0.14 [-0.04 to 0.32]
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; Mean difference between receiving the intervention and not receiving the intervention at each time point; Test type: Superiority; p = 0.13, Regression, Linear; β = 0.14, z = 1.51

6. Secondary Outcome: Average Change in d Score on digiBP From One Decision Time Point to the Next Decision Time Point as a Result of the Intervention
Description: Mood was self-reported using the 6-item digital survey for mood in bipolar disorder (digiPB). This survey is comprised of 3 items (depressed mood, fatigue, fidgeting) measuring common depressive symptoms, two items (increased energy, rapid speech) measuring common manic symptoms, and one item (irritability) measuring a common symptom of both mania and depression. Each item is rated on ordinal scale: 0=absent/normal, 1=mild, 2=moderate, 3=severe. Two scores, d and m, are computed to measure severity of depressive and manic symptoms, respectively. D score ranges from 0 to 21, higher scores being most severe symptoms of depression. Self-reported mood was collected twice-daily over 42 days, once in the morning and once in the evening. This leads to a total of 84 decision time points. This outcome looks at the average change in the d score from one decision time point to the next (e.g., from morning to evening or from evening to the next morning) that is attributed to the intervention.
Time Frame: data collected twice daily over 42 days (Days 1-43)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 26
score on a scale | 0.38 [0.11 to 0.65]
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; Mean difference between receiving the intervention and not receiving the intervention at each time point; Test type: Superiority; p = 0.007, Regression, Linear; β = 0.38, z = 2.71

7. Secondary Outcome: Average Change in Toward Energy Score From One Decision Time Point to the Next Decision Time Point as a Result of the Intervention
Description: The effectiveness of the ACT micro-intervention will be assessed by looking at responses to the activity questionnaire in relation to whether or not a participant received a micro-intervention at the prior time-point.
  Since you [woke this morning or last logged your symptoms], how much energy was consumed by pursuing your values (example: making choices that align with who you want to be or who/what matters)?
  Questions are answered using a scale of 0-6, where 0 = "none" and 6 = "all of my energy."
  Self-reported toward energy was collected twice-daily over 42 days, once in the morning and once in the evening. This leads to a total of 84 decision time points. This outcome looks at the average change in toward energy from one decision time point to the next (e.g., from morning to evening or from evening to the next morning) that is attributed to the intervention.
Time Frame: data collected twice daily over 42 days (Days 1-43)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 26
score on a scale | 0.03 [-0.07 to 0.14]
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; Mean difference between receiving the intervention and not receiving the intervention at each time point; Test type: Superiority; p = 0.57, Regression, Linear; β = 0.03, z = 0.58

8. Secondary Outcome: Average Change in Away Energy Score From One Decision Time Point to the Next Decision Time Point as a Result of the Intervention
Description: The effectiveness of the ACT micro-intervention will be assessed by looking at responses to the activity questionnaire in relation to whether or not a participant received a micro-intervention at the prior time-point.
  Since you [woke this morning or last logged your symptoms], how much energy was consumed by trying to get rid of unwanted feelings, thoughts, or other internal experiences (example: suppressing, distracting, avoiding)?
  Questions are answered using a scale of 0-6, where 0 = "none" and 6 = "all of my energy."
  Self-reported away energy was collected twice-daily over 42 days, once in the morning and once in the evening. This leads to a total of 84 decision time points. This outcome looks at the average change in away energy from one decision time point to the next (e.g., from morning to evening or from evening to the next morning) that is attributed to the intervention.
Time Frame: data collected twice daily over 42 days (Days 1-43)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACT-based Microintervention Delivered by Mobile App
Number analyzed (Participants) | 26
score on a scale | 0.06 [-0.04 to 0.16]
Statistical Analysis 1: Comparison: ACT-based Microintervention Delivered by Mobile App; Mean difference between receiving the intervention and not receiving the intervention at each time point; Test type: Superiority; p = 0.25, Regression, Linear; β = 0.06, z = 1.15

ADVERSE EVENTS:
Time Frame: up to day 42
Description: Other Reportable Incidence or Occurrences (ORIOs) are also reported.
Arm/Group | ACT-based Microintervention Delivered by Mobile App
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-based Microintervention Delivered by Mobile App (N=30)
Sensory Processing Disorder (Nervous system disorders) | 1 (1) — Participant discontinued from the study due to problems with sensory processing disorder. Participant agreed to still complete the final interview.
Fitbit Specific Device Issues (Product Issues) | 9 (9)
Technology Issues (Product Issues) | 5 (5) — Study app troubleshooting or participant problems working with it

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT04098497/Prot_SAP_000.pdf